CLINICAL TRIAL: NCT01369680
Title: Oral Ketamine for Control of Chronic Pain in Children
Acronym: KETA-2011
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, David Korones, Director, Pediatric Palliative Care, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KETA-2011
Record Dates: First submitted 2011-05-23; First posted 2011-06-09 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Pain
Keywords: Ketamine; Chronic pain; Children; Oral pain medication
MeSH Terms: conditions — Chronic Pain | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ketamine 0.25 mg/kg/dose (Experimental): The first three subjects were administered 0.25 mg/kg/dose oral ketamine.
  Interventions: Drug: Ketamine
- Ketamine 0.5 mg/kg/dose (Experimental): The second group of three subjects were administered 0.5 mg/kg/dose oral ketamine.
  Interventions: Drug: Ketamine
- Ketamine 1 mg/kg/dose (Experimental): The third group of three subjects were administered 1 mg/kg/dose oral ketamine.
  Interventions: Drug: Ketamine
- Ketamine 1.5 mg/kg/dose (Experimental): The fourth group of three subjects were administered 1.5 mg/kg/dose oral ketamine.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Drug will be given orally three times a day at doses escalating from 0.25mg/kg/dose to 1.5mg/kg/dose in cohorts of 3. Each subject will be administered study drug for 2 weeks.
  Other Names: Ketalar; Ketamine hydrochloride

SUMMARY:
The study is a maximum tolerated dose finding study for oral, chronic, daily administration of oral ketamine (by mouth) in children with long-term daily pain.

DETAILED DESCRIPTION:
Pain control in children is a major concern when children have chronic diseases, such as cancer and sickle cell disease with frequent pain crises. Additionally, though the traditional pain medications of morphine and acetaminophen are regarded as safe and effective for pain control in children, there are few alternative therapies available when these medications are insufficient. Chronic pain (whether cancer or non-cancer pain) in children has few approved and well tolerated therapeutic options with proven efficacy.

Ketamine is a medication that was first described in 1962[1]. It is an NMDA-R (N-methyl-D-aspartate-receptor) antagonist with dissociative amnestic and analgesic effects[1-2]. Ketamine is particularly successful as a dissociative amnestic for children in the emergent setting as it has little respiratory or cardiac impact, has a short half-life, and has fewer psychomimetic effects in the pediatric population than in adults[1]. Its function is via antagonism and reduction of NMDA-receptors in the afferent pain pathway. In effect, this decreases pain receptors and can dramatically reduce the need for narcotic pain medications for patients with chronic pain.

Unfortunately, with such dissociative effects, ketamine has been a drug of abuse for decades[1,3]. Additionally, there is concern that ketamine may have long-term deleterious effects on cognition for those subjects chronically exposed to IV ketamine[4], especially children whose neural pathways may still be developing[1,5]. These effects may include difficulty with attention and working memory, though the effects appear to be short-term and reversible in adults. However, much of this data is derived from rodent or primate studies, and there is little evidence that there are long-term cognitive effects on humans chronically exposed to ketamine[1]. This lack of data is particularly impactful in the pediatric group.

Ketamine has been evaluated as an analgesic medication for patients with chronic pain that is not resolved with narcotics and gabapentin. There are a number of case reports and small case series that suggest ketamine is a useful medication for control of chronic pain in adults[2,4,6-8]. Additionally, there are case studies that describe lasting (12 week) pain control in adults after 4-10 days of ketamine therapy[7-8]. However, there are, to date, little data that aid a pediatrician in determining if ketamine is a safe and effective option as a chronic, oral therapy for children with chronic pain.

Overall, there are few proven safe and effective medications for use in chronic pain management for children. Ketamine is a well known medication with a well elaborated safety profile, when given intravenously and for short periods of time. There is, as above, emerging data that ketamine is useful for chronic pain control in adults. The question that remains to be answered is whether ketamine is a safe option for chronic use in children, whose brains are significantly more plastic and whose metabolism is different compared with those of adults.

ELIGIBILITY:
Inclusion Criteria:

* Subject, parent, or guardian willing and able to give informed consent
* NRS for pain >4
* Chronic pain, which has been present for >3 months, or persisting longer than is normal for the underlying diagnosis
* Chronic pain related to diagnoses including but not limited to: cancer, rheumatologic disease, sickle cell anemia, cystic fibrosis, pancreatitis, and neuromuscular disease (e.g. Duchenne muscular dystrophy)
* Able to tolerate and cooperate with neurocognitive assessment
* Age 8-22 years old

Exclusion Criteria:

* If they are known or suspected to have drug dependence or addiction
* History of psychiatric disorder such as depression, schizophrenia, or bipolar disorder
* History of hypertension
* Unable to cooperate with neurocognitive assessment
* Chronic pain related to chronic abdominal pain syndrome
* Known liver disease or elevation of AST or ALT greater than 3 times the upper limit of normal.
* Previous intolerance or allergic reaction to ketamine
* Pregnancy
* Use of CYP3A4 inhibitors or inducers within the 2 week period prior the study drug administration or within 5 half-lives of the respective medication, whichever is longer, until study conclusion.
* Consumption of grapefruit or grapefruit products from at least 2 weeks prior to study drug administration until study conclusion.

Ages: 8 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Korones, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Green SM, Cote CJ. Ketamine and neurotoxicity: clinical perspectives and implications for emergency medicine. Ann Emerg Med. 2009 Aug;54(2):181-90. doi: 10.1016/j.annemergmed.2008.10.003. Epub 2008 Nov 6. PMID 18990467
- [Background] Okon T. Ketamine: an introduction for the pain and palliative medicine physician. Pain Physician. 2007 May;10(3):493-500. PMID 17525784
- [Background] Kronenberg RH. Ketamine as an analgesic: parenteral, oral, rectal, subcutaneous, transdermal and intranasal administration. J Pain Palliat Care Pharmacother. 2002;16(3):27-35. doi: 10.1080/j354v16n03_03. PMID 14640353
- [Background] Visser E, Schug SA. The role of ketamine in pain management. Biomed Pharmacother. 2006 Aug;60(7):341-8. doi: 10.1016/j.biopha.2006.06.021. Epub 2006 Jul 5. PMID 16854557
- [Background] Wilder RT, Flick RP, Sprung J, Katusic SK, Barbaresi WJ, Mickelson C, Gleich SJ, Schroeder DR, Weaver AL, Warner DO. Early exposure to anesthesia and learning disabilities in a population-based birth cohort. Anesthesiology. 2009 Apr;110(4):796-804. doi: 10.1097/01.anes.0000344728.34332.5d. PMID 19293700
- [Background] Schwartzman RJ, Alexander GM, Grothusen JR, Paylor T, Reichenberger E, Perreault M. Outpatient intravenous ketamine for the treatment of complex regional pain syndrome: a double-blind placebo controlled study. Pain. 2009 Dec 15;147(1-3):107-15. doi: 10.1016/j.pain.2009.08.015. Epub 2009 Sep 23. PMID 19783371
- [Background] Sigtermans MJ, van Hilten JJ, Bauer MCR, Arbous SM, Marinus J, Sarton EY, Dahan A. Ketamine produces effective and long-term pain relief in patients with Complex Regional Pain Syndrome Type 1. Pain. 2009 Oct;145(3):304-311. doi: 10.1016/j.pain.2009.06.023. Epub 2009 Jul 14. PMID 19604642
- [Background] Bell RF. Ketamine for chronic non-cancer pain. Pain. 2009 Feb;141(3):210-214. doi: 10.1016/j.pain.2008.12.003. Epub 2009 Jan 6. No abstract available. PMID 19128879
- [Derived] Bredlau AL, McDermott MP, Adams HR, Dworkin RH, Venuto C, Fisher SG, Dolan JG, Korones DN. Oral ketamine for children with chronic pain: a pilot phase 1 study. J Pediatr. 2013 Jul;163(1):194-200.e1. doi: 10.1016/j.jpeds.2012.12.077. Epub 2013 Feb 10. PMID 23403253

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in June 2011 and closed in April 2012. Patients were referred by their primary pain physician.
Groups:
- Ketamine 0.25 mg/kg/Dose: Cohort of three participants treated at 0.25 mg/kg/dose oral ketamine.
- Ketamine 0.5 mg/kg/Dose: Cohort of three participants treated at 0.5 mg/kg/dose oral ketamine.
- Ketamine 1 mg/kg/Dose: Cohort of three participants treated at 1 mg/kg/dose oral ketamine.
- Ketamine 1.5 mg/kg/Dose: Cohort of three participants treated at 1.5 mg/kg/dose oral ketamine.
Period: Overall Study
Arm/Group | Ketamine 0.25 mg/kg/Dose | Ketamine 0.5 mg/kg/Dose | Ketamine 1 mg/kg/Dose | Ketamine 1.5 mg/kg/Dose
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 2 | 1
Not Completed | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine 0.25 mg/kg/Dose | Ketamine 0.5 mg/kg/Dose | Ketamine 1 mg/kg/Dose | Ketamine 1.5 mg/kg/Dose | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 3 | 3 | 3 | 11
  Between 18 and 65 years | 1 | 0 | 0 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 1 | 9
  Male | 0 | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Tolerating Dose
Description: According to CTCae any dose causing grade 2 or worse toxicity will be an untolerated dose. Tolerability is defined as ability to take the medication for 2 weeks without having a grade 2 or worse toxicity.
Time Frame: Up to 2 weeks
Population: Number of participants was determined through negotiation with the FDA for safety of all participants.
Measure: Number; unit: participants
Groups:
- Ketamine 0.25 mg/kg/Dose: Cohort of three subjects administered 0.25 mg/kg/dose oral ketamine
- Ketamine 0.5 mg/kg/Dose: Cohort of three subjects administered 0.5 mg/kg/dose oral ketamine
- Ketamine 1 mg/kg/Dose: Cohort of three subjects administered 1 mg/kg/dose oral ketamine
- Ketamine 1.5 mg/kg/Dose: Cohort of three subjects administered 1.5 mg/kg/dose oral ketamine
Arm/Group | Ketamine 0.25 mg/kg/Dose | Ketamine 0.5 mg/kg/Dose | Ketamine 1 mg/kg/Dose | Ketamine 1.5 mg/kg/Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3
participants | 3 | 3 | 3 | 1

2. Secondary Outcome: Neurocognitive Effect
Description: Baseline neurocognitive testing will be done before study drug is given. Subjects will be reassessed for any changes in neurocognitive scores at end of dosing (week 2) and at three weeks off study drug (week 14). Significant changes were measured at week 14 compared to baseline. Week 2 was measured to inform future studies.
  The neurocognitive scores are standardized scores with a mean of 100; low scores correlate with low neurocognitive function, while high scores correlate with high function. A significant change is defined as greater than or equal to 10% decrease in scores.
Time Frame: At 14 weeks
Population: All participants not lost to follow-up were analyzed
Measure: Number; unit: participants
Groups:
- Ketamine 0.25 mg/kg/Dose: Cohort of three subjects administered 0.25 mg/kg/dose oral ketamine. Measure was for clinically significant decline in neurocognitive scores.
- Ketamine 0.5 mg/kg/Dose: Cohort of three subjects administered 0.5 mg/kg/dose oral ketamine. Measure was for clinically significant decline in neurocognitive scores.
- Ketamine 1 mg/kg/Dose: Cohort of three subjects administered 1 mg/kg/dose oral ketamine. Measure was for clinically significant decline in neurocognitive scores.
- Ketamine 1.5 mg/kg/Dose: Cohort of three subjects administered 1.5 mg/kg/dose oral ketamine. Measure was for clinically significant decline in neurocognitive scores.
Arm/Group | Ketamine 0.25 mg/kg/Dose | Ketamine 0.5 mg/kg/Dose | Ketamine 1 mg/kg/Dose | Ketamine 1.5 mg/kg/Dose
Number analyzed (Participants) | 3 | 3 | 2 | 1
participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Norketamine Cmax (Measured in ng/mL).
Description: Pharmacokinetic testing will be done during chronic ketamine administration on subjects consenting to additional testing one week into study drug administration. This is to further describe the activity of ketamine in the blood of children when administered chronically and to enable comparison of any clinical effect or toxicity with steady state levels of ketamine in children.
Time Frame: At week 1
Population: All participants consenting for pharmacokinetics were analyzed. No participants in ketamine 1.5 mg/kg/dose group consented for pharmacokinetics.
Measure: Mean (Full Range); unit: ng/mL
Groups:
- Ketamine 0.25 mg/kg/Dose: Subjects treated at 0.25 mg/kg/dose consenting for separate pharmacokinetics test at week 1 of study.
- Ketamine 0.5 mg/kg/Dose: Subjects treated at 0.5 mg/kg/dose consenting for separate pharmacokinetics test at week 1 of study.
- Ketamine 1 mg/kg/Dose: Subjects treated at 1 mg/kg/dose consenting for separate pharmacokinetics test at week 1 of study.
Arm/Group | Ketamine 0.25 mg/kg/Dose | Ketamine 0.5 mg/kg/Dose | Ketamine 1 mg/kg/Dose
Number analyzed (Participants) | 2 | 2 | 1
ng/mL | 37.5 [20 to 55] | 135 [120 to 150] | 250 [250 to 250]

4. Secondary Outcome: Pain Control
Description: Subjects will be assessed for clinically significant change in pain scores during and after study drug administration. Significant change in pain scores were determined at week 2, though week 14 scores were collected as well.
  Participants with a 2 point (or greater) decrease in pain scores compared to baseline were considered to have responded. The NRS scale was used, the scale ranges from 0-10, with 10 being the most pain.
Time Frame: Week 2
Population: Number of participants for analysis was determined in negotiation with the FDA for safety of all participants.
Measure: Number; unit: participants
Groups:
- Ketamine 1 mg/kg/Dose: Cohort of three subjects administered 0.25 mg/kg/dose oral ketamine.
Arm/Group | Ketamine 0.25 mg/kg/Dose | Ketamine 0.5 mg/kg/Dose | Ketamine 1 mg/kg/Dose | Ketamine 1.5 mg/kg/Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3
participants | 3 | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Ketamine 0.25 mg/kg/Dose | Ketamine 0.5 mg/kg/Dose | Ketamine 1 mg/kg/Dose | Ketamine 1.5 mg/kg/Dose
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine 0.25 mg/kg/Dose (N=3) | Ketamine 0.5 mg/kg/Dose (N=3) | Ketamine 1 mg/kg/Dose (N=3) | Ketamine 1.5 mg/kg/Dose (N=3)
Infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) — Multiple infections in one subject with complex medical diagnoses. Not thought to be related to study drug.
Pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine 0.25 mg/kg/Dose (N=3) | Ketamine 0.5 mg/kg/Dose (N=3) | Ketamine 1 mg/kg/Dose (N=3) | Ketamine 1.5 mg/kg/Dose (N=3)
Confusion (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Withdrawal from chronic opioid therapy.
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pain (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Relieved with defecation
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Three subjects were lost to follow-up, limiting the data available for neuro-cognitive assessment at the last visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No